CLINICAL TRIAL: NCT05401136
Title: Evaluating the Hepatitis C Chain of Addiction Care Pathway for People Who Inject(ed) Drugs in Addiction Care
Brief Title: Evaluating the Chain of Addiction Care (CAC)
Acronym: HepC:CAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: AbbVie (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-5939
Record Dates: First submitted 2022-05-24; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C, Chronic; Substance Use Disorders
MeSH Terms: conditions — Hepatitis C, Chronic; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Consecutive people who use drugs and visit the addiction care centre

SUMMARY:
The investigators want to evaluate the feasibility of a decentralised hepatitis C care pathway (the Chain of Addiction Care (CAC) pathway) in several addiction care centres in the east of the Netherlands. Secondary objective: to measure the impact of hepatitis C clearance on MET (+metabolite) and BUP (+metabolite) trough levels in patients on Opioid substitution Therapy (OST). This is an exploratory, observational study.

DETAILED DESCRIPTION:
People who (have) inject(ed) drugs (PWID) are at high risk for hepatitis C infection. Establishing adequate linkage to care in this population can be a challenge. Many of these patients receive opioid substitution, hepatitis C treatment possibly influences pharmacokinetics of those substitutes. This protocol describes a study on hepatitis C in people who (have) inject(ed) drugs (PWID), consisting of two substudies. 1) An exploratory, observational study in which we evaluate the decentralised hepatitis C care pathway in addiction care centres. 2) An observational pharmacokinetic study in hepatitis C patients on opioid substitution therapy (OST) embedded within the first study.

Rationale: 1) Many PWIDs are lost during the process of testing and linkage to care and do therefore not receive adequate hepatitis C treatment. Decentralising care in addiction care centres deems hospital visits unnecessary, an approach that has become increasingly popular in this population over the last few years. This practice however has not yet been evaluated in the Netherlands. 2) In the Netherlands the PWID population is often treated for opioid addiction by opioid substitution therapy (OST) with methadone (MET) or buprenorphine (BUP). There is evidence that liver inflammation has a negative effect on pharmacokinetics of drugs. Consequently, we hypothesize that HCV treatment results in reduced liver inflammation and a decrease in MET and/or BUP levels, which is clinically relevant in the PWID/OST population.

Objective: 1) to evaluate the feasibility of a decentralised hepatitis C care pathway (the Chain of Addiction Care (CAC) pathway) in several addiction care centres in the east of the Netherlands. 2. to measure the impact of hepatitis C clearance on MET (+metabolites) and BUP (+metabolites) levels and craving in patients on OST.

Study design: This is an exploratory, observational study with a pharmacokinetic observational study embedded within the same population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able and willing to give informed consent
* Currently inject or previously injected drugs at least once, including nasal snorting of drugs using aids such as basepipes or straws.
* Visit the participating addiction care centre at least once during the study period

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PWID of 18 years or older who visit the participating addiction care centre
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
HCV prevalence (both anti-HCV and HCV RNA). | At screening (week 0)
  Participants are invited to undergo viral hepatitis screening (standard care)
Treatment acceptance rate. | After evaluation (~week 3)
  Participants with chronic HCV infection are invited to be treated (standard care)
Sustained virologic response | 12 weeks after treatment (~week 30)
  Participants who were treated and were 'cured' (standard care)

SECONDARY OUTCOMES:
Acceptance rate of on-site testing. | through study completion, an average of 1 year
  Number of participants that engage in testing
Re-infection rate. | through study completion, an average of 1 year
  Patients re-infected after successful treatment
Mean decrease in MET and BUP trough levels | through study completion, an average of 1 year
  Difference in concentration of methadone or buprenorphine before and after treatment.
Change in dosage of MET and BUP during follow-up | through study completion, an average of 1 year
  Physician initiated dosage change before compared to after treatment of hepatitis C
Patient reported drug use | through study completion, an average of 1 year
  Drug use during study timeframe

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Von den Hoff DW, Berden FAC, Drenth JPH, Schellekens AFA; HepNed, NISPA. Implementation of a decentralized hepatitis C care pathway for people who use drugs in Dutch addiction care. Study protocol for the Hepatitis C: chain of addiction care (CAC) project. Addict Sci Clin Pract. 2022 Nov 30;17(1):67. doi: 10.1186/s13722-022-00350-1. PMID 36451175